CLINICAL TRIAL: NCT02299713
Title: Randomized, Double-Blind, Placebo-Controlled Trial, Parallel Design Used To Evaluate Pain, Endocrinologic Variations, Life Quality And Medication Use, After Electro-Acupuncture Treatment In Patients With Osteoarthritis Of The Knee
Brief Title: Electro-Acupuncture Treatment in Patients With Osteoarthritis Of The Knee (EATOAK)
Acronym: EATOAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Son Llatzer (Other)
Responsible Party: Principal Investigator, Javier Mata, Chief of Section of Anesthesiology and Reanimation Department, Hospital Son Llatzer
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ACU-001
Record Dates: First submitted 2014-11-11; First posted 2014-11-24 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis, Knee
Keywords: acupuncture; knee pain
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo/sham acupuncture (Sham Comparator): There are different types of controls used in acupuncture trials. We used the control described as sham and by some as minimal acupuncture. This group had the same schedule as the electro-acupuncture group. Sham acupuncture was administered, with the same duration and frequency and by the same specialist who performed the non-sham acupuncture. Retractable needles were placed into small adhesive cylinders, so that the needles were supported but did not perforate the skin. The acupuncturist placed the needles at the same points as the non-sham group and used the same pairs of electrodes to simulate the electrical connection.
  Interventions: Device: Electroacupuncture
- Electroacupuncture (Active Comparator): The electro-acupuncture device was a biphasic pulse generator. It was used with maximum tolerable intensity of current and a frequency of 3 Hz. The points were selected according to the Traditional Chinese Medicine meridian theory to treat knee pain. The points selected were local points St 34, St 35, St 36,Liv 8, Sp 10. One distal point St 44.A total of six needles were inserted into each leg by the acupuncturist (the out come measures were not specifically targeted to whether the patient had one or both knees involved). All patients belonging to this group experienced a De Qi sensation, which is a tingling and numbness sensation upon needling of specific points.
  Interventions: Device: Electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture — Electro acupuncture is a relatively new method of treatment in Chinese Medicine. Just as in a regular acupuncture treatment, needles are inserted into acupuncture points but small crocodile clips are then attached to the ends of needles to connect them to an electro-acupuncture device. In traditional acupuncture the inserted needles are manually vibrated to induce a response whilst in electro-acupuncture the bi-phasic current results in a constant (controlled) vibration of the needles and a direct electrical stimulation. The device allows the practitioner to adjust the frequency and intensity of the electric stimulation in a consistent manner which is not operator dependant.

SUMMARY:
The purpose of this study is to assess the efficacy of electroacupuncture (EA) on pain control, perception of pain, plasma cortisol and beta-endorphins levels, patient-perceived quality of life and use of pain medications, in people with chronic knee pain.

DETAILED DESCRIPTION:
Previous randomised trials and meta-analyses have shown certain efficacy of acupuncture in some chronic painful conditions, in spite of methodological weaknesses. The hypothalamic-pituitary-adrenal (HPA) axis and the endogenous opioid (EO) system are the mechanisms appear to explain how acupuncture works in part. These systems have been shown to be important mediators of stress, pain and other stimuli. The Osteoarthritis Research International suggest that osteoarthritis (OA) treatment should be multidisciplinary and recommended acupuncture as one of 12 possible non-pharmacological modalities for treating OA.

This study is a randomized, double-blind, placebo-controlled trial, parallel design. 128 out-patients over 50 years with OA of the knee will be recruited from Mallorca, Spain. Participants will be randomly allocated into two groups: placebo/sham acupuncture, non insertion technique, and EA. Acupuncture treatments will be used the Traditional Chinese Medicine (TCM) style. The patients will be evaluated after a period of one month (2 sessions weekly), three months (1session monthly), six months (1 session every 45 days) and again one year later (1 session every 2 months), at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex with primary osteoarthritis of one or both knees fulfilling diagnostic criteria for osteoarthritis knee laid down by American College of Rheumatology.
* Patients also had to have a Kellgren-Lawrence (radiologic criterion) score of at least 2 and chronic pain in the knee joint for more than 3 months.

Exclusion Criteria:

* The patients with secondary osteoarthritis of knees
* Associated systemic arthropathies, e.g. rheumatoid arthritis and gout
* Patients on steroids
* Disease modifying drugs, e.g. methotrexate and azathioprine
* Patients with recent trauma in the area of acupuncture
* History of intra articular injection of steroid within last two months
* Patients missing two or more sessions of electro-acupuncture consecutively were excluded from the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-01; Primary Completion 2017-02 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in visual analogue scale (VAS) and the Western Ontario and McMaster (WOMAC) Universities Osteoarthritis Index pain subscale | baseline and the completion of treatment at 12 weeks.
  a continuous scale comprised of a horizontal line, anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale]). (VAS pain intensity score)

SECONDARY OUTCOMES:
Changes from baseline in The Short Form 36 version 2 (SF-36v2) health survey | at 1 month
  patient-perceived quality of life
Changes from baseline in The Short Form 36 version 2 (SF-36v2) health survey | at 3 months
  patient-perceived quality of life
Changes from baseline in The Short Form 36 version 2 (SF-36v2) health survey | at 6 months
  patient-perceived quality of life
Changes from baseline in The Short Form 36 version 2 (SF-36v2) health survey | up to 1 year
  patient-perceived quality of life
Change from baseline in plasma cortisol and beta-endorphins levels | at 1 month
  analysis of blood samples
Change from baseline in plasma cortisol and beta-endorphins levels | at 3 months
  analysis of blood samples
Change from baseline in plasma cortisol and beta-endorphins levels | at 6 months
  analysis of blood samples
Change from baseline in plasma cortisol and beta-endorphins levels | up to 1 year
  analysis of blood samples
Change from Baseline in Goldberg Depression and Anxiety scales | at 1 month
  measured with the Goldberg Anxiety and Depression Scale. The Spanish version validated by Montón et al. will be used
Change from Baseline in Goldberg Depression and Anxiety scales | at 3 months
  measured with the Goldberg Anxiety and Depression Scale. The Spanish version validated by Montón et al. will be used
Change from Baseline in Goldberg Depression and Anxiety scales | at 6 months
  measured with the Goldberg Anxiety and Depression Scale. The Spanish version validated by Montón et al. will be used
Change from Baseline in Goldberg Depression and Anxiety scales | up to 1 year
  measured with the Goldberg Anxiety and Depression Scale. The Spanish version validated by Montón et al. will be used
Change from baseline in WOMAC index | at 1 month
  WOMAC scale. There are two questions for stiffness (scale of 0-8) and 17 questions for functional limitation (score range of 0-68). Each question will be answered orally with the following criteria: "none" = 0, "a bit" = 1, "quite a bit" = 2, "a lot" = 3, and "very much" = 4. If two or more questions are unanswered, the scale scores will be declared invalid and not counted.
Change from baseline in WOMAC index | at 6 months
  WOMAC scale. There are two questions for stiffness (scale of 0-8) and 17 questions for functional limitation (score range of 0-68). Each question will be answered orally with the following criteria: "none" = 0, "a bit" = 1, "quite a bit" = 2, "a lot" = 3, and "very much" = 4. If two or more questions are unanswered, the scale scores will be declared invalid and not counted.
Change from baseline in WOMAC index | up to 1 year
  WOMAC scale. There are two questions for stiffness (scale of 0-8) and 17 questions for functional limitation (score range of 0-68). Each question will be answered orally with the following criteria: "none" = 0, "a bit" = 1, "quite a bit" = 2, "a lot" = 3, and "very much" = 4. If two or more questions are unanswered, the scale scores will be declared invalid and not counted.
Changes in baseline use of medication | at 1 month
  EUROHIS (European Health Survey System) theoretical recommendations and design of a questionnaire
Changes in baseline use of medication | at 3 months
  EUROHIS (European Health Survey System) theoretical recommendations and design of a questionnaire
Changes in baseline use of medication | at 6 months
  EUROHIS (European Health Survey System) theoretical recommendations and design of a questionnaire
Changes in baseline use of medication | up to 1 year
  EUROHIS (European Health Survey System) theoretical recommendations and design of a questionnaire
Change from baseline in a visual analogue scale (VAS) | at 1 month
  a continuous scale comprised of a horizontal line, anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale]). (VAS pain intensity score)
Change from baseline in a visual analogue scale (VAS) | at 6 months
  a continuous scale comprised of a horizontal line, anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale]). (VAS pain intensity score)
Change from baseline in a visual analogue scale (VAS) | up to 1 year
  a continuous scale comprised of a horizontal line, anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale]). (VAS pain intensity score)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Mata, M.D., Principal Investigator — Anaesthesia Department, Son Llàtzer University Hospital. Palma de Mallorca. Spain
Locations (2):
- Spain (2):
  - Son Llatzer University Hospital, Palma, Balear Islands
  - Son LLàtzer Hospital, Palma, Balearic Islands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahsin S, Saleem S, Bhatti AM, Iles RK, Aslam M. Clinical and endocrinological changes after electro-acupuncture treatment in patients with osteoarthritis of the knee. Pain. 2009 Dec 15;147(1-3):60-6. doi: 10.1016/j.pain.2009.08.004. Epub 2009 Sep 18. PMID 19766392
- [Background] Vas J, Mendez C, Perea-Milla E, Vega E, Panadero MD, Leon JM, Borge MA, Gaspar O, Sanchez-Rodriguez F, Aguilar I, Jurado R. Acupuncture as a complementary therapy to the pharmacological treatment of osteoarthritis of the knee: randomised controlled trial. BMJ. 2004 Nov 20;329(7476):1216. doi: 10.1136/bmj.38238.601447.3A. Epub 2004 Oct 19. PMID 15494348
- [Background] Sangdee C, Teekachunhatean S, Sananpanich K, Sugandhavesa N, Chiewchantanakit S, Pojchamarnwiputh S, Jayasvasti S. Electroacupuncture versus diclofenac in symptomatic treatment of osteoarthritis of the knee: a randomized controlled trial. BMC Complement Altern Med. 2002 Mar 21;2:3. doi: 10.1186/1472-6882-2-3. PMID 11914160
- [Background] Witt C, Brinkhaus B, Jena S, Linde K, Streng A, Wagenpfeil S, Hummelsberger J, Walther HU, Melchart D, Willich SN. Acupuncture in patients with osteoarthritis of the knee: a randomised trial. Lancet. 2005 Jul 9-15;366(9480):136-43. doi: 10.1016/S0140-6736(05)66871-7. PMID 16005336
- [Background] Berman BM, Lao L, Langenberg P, Lee WL, Gilpin AM, Hochberg MC. Effectiveness of acupuncture as adjunctive therapy in osteoarthritis of the knee: a randomized, controlled trial. Ann Intern Med. 2004 Dec 21;141(12):901-10. doi: 10.7326/0003-4819-141-12-200412210-00006. PMID 15611487
- [Background] Selfe TK, Taylor AG. Acupuncture and osteoarthritis of the knee: a review of randomized, controlled trials. Fam Community Health. 2008 Jul-Sep;31(3):247-54. doi: 10.1097/01.FCH.0000324482.78577.0f. PMID 18552606
- [Background] Kwon YD, Pittler MH, Ernst E. Acupuncture for peripheral joint osteoarthritis: a systematic review and meta-analysis. Rheumatology (Oxford). 2006 Nov;45(11):1331-7. doi: 10.1093/rheumatology/kel207. Epub 2006 Aug 27. PMID 16936326
- [Background] White A, Foster NE, Cummings M, Barlas P. Acupuncture treatment for chronic knee pain: a systematic review. Rheumatology (Oxford). 2007 Mar;46(3):384-90. doi: 10.1093/rheumatology/kel413. Epub 2007 Jan 10. PMID 17215263
- [Background] Manheimer E, Cheng K, Linde K, Lao L, Yoo J, Wieland S, van der Windt DA, Berman BM, Bouter LM. Acupuncture for peripheral joint osteoarthritis. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD001977. doi: 10.1002/14651858.CD001977.pub2. PMID 20091527
- [Derived] Mata J, Cabrera S, Sanchis P, Valenti P, Hernandez P, Fortuny R, Lirola S, Aguilar JL. Electro-acupuncture for treatment of knee pain from osteoarthritis and the possible endocrinology changes: a study protocol for a randomized controlled trial. Trials. 2015 Jun 3;16:248. doi: 10.1186/s13063-015-0766-2. PMID 26037626